CLINICAL TRIAL: NCT06494228
Title: Comparison of Diagnostic Performances of 3D FLAIR, DIR and PSIR Sequences in Optic Neuritis
Acronym: Optic-Neuritis
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9024
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis; Demyelinating Diseases
Keywords: Multiple Sclerosis; Demyelinating Diseases
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ultimately improve the care of patients suffering from multiple sclerosis (1st cause of acquired non-traumatic disability in adults) and NMO spectrum diseases by using more efficient MRI sequences than the FLAIR sequence commonly used in detection of optic neuritis.

In the literature, many studies have already focused on comparing the sensitivity of detection of white matter demyelination plaques using FLAIR, PSIR or DIR sequences.

Some authors have shown better sensitivity of the PSIR sequence in the detection of demyelinating lesions of the marrow in multiple sclerosis compared to conventional sequences.

Others have shown better performance of the combined use of PSIR and DIR sequences compared to the FLAIR sequence in the detection of cortical lesions in multiple sclerosis.

However, in the context of optic neuritis, few comparative studies comparing these three sequences have been carried out:

A 2022 study showed better diagnostic sensitivity of optic neuritis of the DIR sequence compared to the FLAIR sequence.

A possible better diagnostic performance of a sequence not used in current practice in the detection of optic neuritis (PSIR and DIR sequences), would be possible to justify their use on a larger scale and ultimately improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject suffering from multiple sclerosis or an NMO spectrum disease
* Subject having received an MRI including 3D FLAIR, 3D DIR and 3D PSIR sequences
* Brain MRIs of eligible subjects acquired between April 1, 2019 and November 30, 2021.
* No opposition to the reuse of its data for scientific research purposes.

Exclusion Criteria:

* Presence of opposition from the subject (and/or their legal representative if applicable) to the reuse of their data for scientific research purposes.
* Artifacts not allowing satisfactory interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥18 years old), suffering from multiple sclerosis or an NMO spectrum disease, and having received an MRI including 3D FLAIR, 3D DIR and 3D PSIR sequences between April 1, 2019 and November 30 2021.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01-19 (Estimated)

PRIMARY OUTCOMES:
Comparison of the radiologist's degree of diagnostic confidence based on the three sequences (3D FLAIR, 3D DIR and 3D PSIR sequences). | One month after brain MRI
  During their analysis, each investigator fills out an interpretation grid for each series, where they indicate the presence or absence of optic neuritis and the degree of confidence they attribute to it on a scale of 1 to 5.
  During their analysis, each investigator fills out an interpretation grid for each series, where they indicate the presence or absence of optic neuritis and the degree of confidence they attribute to it on a scale of 1 to 5.
  A score of 5 shows that the level of confidence is very good.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie II, CHU de Strasbourg, Strasbourg, Les Hôpitaux Universitaires de Strasbourg, France